CLINICAL TRIAL: NCT02254655
Title: The Effect of Puerarin Injection on Carotid Intima-Media Thickness in Patients With Rheumatoid Arthritis, a Controlled and Randomized Trial
Brief Title: The Effect of Puerarin Injection on Carotid Intima-Media Thickness in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yang Min, Dr., Chengdu PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-2012-063; No. BWS11J067 (Other Grant/Funding Number: Scientific Research Funds Project of Chinese PLA)
Record Dates: First submitted 2013-11-18; First posted 2014-10-02 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Rheumatoid Arthritis
Keywords: puerarin; rheumatoid arthritis; atherosclerosis; carotid intima-media thickness
MeSH Terms: conditions — Arthritis, Rheumatoid; Atherosclerosis | interventions — puerarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Puerarin injection 400 mg (Experimental): Patients were administrated with 400 mg intravenously infused puerarin injection once a day. Puerarin injection was prepared in 250 mL 0.9% sodium chloride injection before the use. The treatment course consisted of 2 weeks followed by a 15-day interval for 24 weeks. Furthermore, patients receive stable treatment with oral anti-rheumatic agents and/or non-steroidal anti-inflammatory drugs, prednisone, aspirin, statins, bone metabolism regulators and gastric mucosal protective agents on as-needed basis.
  Interventions: Drug: Puerarin injection 400 mg
- Control (Sham Comparator): Patients receive routine anti-rheumatic care only. Patients receive stable treatment with oral anti-rheumatic agents and/or non-steroidal anti-inflammatory drugs, prednisone, aspirin, statins, bone metabolism regulators and gastric mucosal protective agents on as-needed basis.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Puerarin injection 400 mg — Patients receive treatment with oral anti-rheumatic agents and/or non-steroidal anti-inflammatory drugs, prednisone, aspirin, statins, bone metabolism regulators and gastric mucosal protective agents on as-needed basis.Furthermore, patients were administrated with 400 mg intravenously infused puerarin injection once a day.Each treatment course lasted for 2 weeks followed by a regular time interval of 15 days.
  Other Names: Puerarin injection 400 mg + routine anti-rheumatic drugs
  Arms: Puerarin injection 400 mg
Drug: Control — Patients receive treatment with oral anti-rheumatic agents and/or non-steroidal anti-inflammatory drugs, prednisone, aspirin, statins, bone metabolism regulators and gastric mucosal protective agents on as-needed basis
  Other Names: Routine anti-rheumatic drugs
  Arms: Control

SUMMARY:
The purpose of this study is to access the effect (week 12/week 24) of puerarin injection on carotid intima-media thickness (CIMT) in rheumatoid arthritis (RA) patients despite routine anti-rheumatic treatment.

DETAILED DESCRIPTION:
* Controlled, randomized trial
* RA patients under routine anti-rheumatic care were randomized to receive the treatment with or without 400 mg puerarin injection
* Assessments were made at entry, 12 and 24 weeks
* The overall sample size was assessed before the enrollment
* Randomization was performed using concealed random allocation method
* The collected data was processed and assessed by two reviewers
* All the measurement and analysis procedures concerning CIMT were performed by a single ultra sonographer and a single reader, who were blinded to patient profiles and group assignment
* The reproducibility of the ultrasonographic method was test before the trial

ELIGIBILITY:
Inclusion Criteria:

* patients with a definite diagnose of rheumatoid arthritis(RA) were included if they met the classification criteria for RA established by the American Rheumatism Association (ACR) and European League Against Rheumatism (EULAR) in 2010
* aged from 18 to 75 years
* without conflict to the written, informed consent signed prior to the enrollment
* no severe hepatic or renal disorders
* no known carotid artery stenosis
* no coagulation disorders
* no hypertension

Exclusion Criteria:

* being in pregnancy, lactation period or under a pregnancy plan
* being allergic to the test drug
* not compatible for the trial medication
* without full legal capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Carotid intima-media thickness at 24 weeks | At 0 week, 12 weeks, 24 weeks
  Carotid intima-media thickness (CIMT) was using a high-resolution B-mode ultrasound machine (iU22 xMATRIX, Philips, Germany). CIMT was measured twice by a single experienced operator using an 10-MHz linear vascular probe. Patients were let resting in a relaxed supine position, with the head turned gently to the contralateral side when the electrocardiogram was recorded. The imaging system (QLab 6.0, Philips, Germany) was applied to measure the CIMT signals from the proximal internal carotid artery (the arterial segment 10 mm distal to the carotid bifurcation), the carotid bulb and the distal common carotid artery (the arterial segment 10 mm proximal to the carotid bulb). The mean CIMT was calculated from the value of five arterial segments. All the measurement and analysis procedures were performed by a single ultra sonographer and a single reader, who were blinded to patient profiles and group assignment.

SECONDARY OUTCOMES:
low-density lipoprotein cholesterol (LDL-C) | at 0 week, 12 weeks, 24 weeks
erythrocyte sedimentation rate (ESR) | at 0 week, 12 weeks, 24 weeks
C reactive protein (CRP) | at 0 week, 12 weeks, 24 weeks
Total cholesterol (TC) | at 0 week, 12 weeks, 24 weeks
triglycerides (TGs) | at 0 week, 12 weeks, 24 weeks
tumor necrosis factor (TNFα) | at 0 week，12 weeks, 24 weeks
interleukin-8 (IL-8) | at 0 week，12 weeks, 24 weeks
interleukin-1 (IL-1) | at 0 week，12 weeks, 24 weeks
interleukin-6 (IL-6) | at 0 week，12 weeks, 24 weeks
disease activity score in 28 joints (DAS28) | at 0 week，12 weeks, 24 weeks
homeostasis model assessment (HOMA-IR) | at 0 week，12 weeks, 24 weeks

OTHER OUTCOMES:
Kidney function | at 0 week, 12 weeks, 24 weeks
  from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 weeks
Liver function | at 0 week, 12 weeks, 24 weeks
  from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 weeks
blood cell count | at 0 week, 12 weeks, 24 weeks
  from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Min Yang, Ph.D., Principal Investigator — General Hospital of Chengdu Military Area Command PLA

REFERENCES:
- [Derived] Yang M, Luo Y, Liu T, Zhong X, Yan J, Huang Q, Tao J, He Q, Guo M, Hu Y. The Effect of Puerarin on Carotid Intima-media Thickness in Patients With Active Rheumatoid Arthritis: ARandomized Controlled Trial. Clin Ther. 2018 Oct;40(10):1752-1764.e1. doi: 10.1016/j.clinthera.2018.08.014. Epub 2018 Sep 21. PMID 30245282